CLINICAL TRIAL: NCT03178279
Title: An Evaluation of the Use of a Physical Health Plan With People With Psychosis
Brief Title: The Evaluation of the Use of a New Physical Health Plan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRAS194626
Record Dates: First submitted 2017-06-01; First posted 2017-06-06 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2019-10

CONDITIONS: Psychosis; Schizophrenia
Keywords: physical health
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Intervention Model Description: The study will take place in 2 community mental health teams and have 3 main stages. Stage 1: The investigators will undertake focus groups with service users and staff to test out the assumptions in the Theory of Change. Stage 2: The PHP will be available as a paper version and on iPad and smartphone. Each team will be asked to work with all of the people on their caseload to complete the PHP. Service users will be encouraged to complete the PHP whilst waiting for their appointment with their care co-ordinator. The completed PHP will then be emailed to the service user and to their care co-ordinator and they will then be asked to develop an action plan to address any gaps in the completed PHP. Each action plan and the progress made with the action plan will be recorded. This exploratory trial will last six months. Stage 3 The investigators will evaluate the experience of using the PHP using interviews with a random selection of service users and clinical staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of the Physical Health Plan (Experimental): Use of the Physical Health Plan
  Interventions: Other: Physical Health Plan

INTERVENTIONS:
Other: Physical Health Plan — Use of a Physical Health Plan by service users

SUMMARY:
People suffering from psychotic illnesses (e.g. schizophrenia) have poorer physical health than the general population. The reasons include a lack of service user motivation to attend physical health checks and the tendency of health professionals to focus mainly on the mental disorder thus delaying the detection of physical health conditions.

Identifying people who have physical health needs is increasingly recognised as a priority. The investigators have developed a Physical Health Plan (PHP) which is completed by service users and identifies areas of physical health need. An action plan is then completed by the service user and care co-ordinator to address these issues.

The PHP is designed to be very simple to use and there will be 3 versions, 1. paper version, 2. 1 version implemented via the 'IMPARTS' computerised 'tablet' based system that has been separately evaluated (REC Ref 12/SC/0422) and 3. 1 version on an iPad via the MHL2 system via Mindwaves.

The investigators wish to pilot the use of this PHP in two community teams in the South London and Maudsley (SLaM) Trust. The pilot will be done in three stages.

Stage One: The investigators will undertake an initial qualitative study to refine the process of using the PHP using focus group consultations with staff and service users.

Stage Two: The investigators will then undertake a six month study to evaluate the uptake and use of the PHP. This will involve collecting data on how many people complete the PHP and what actions are taken following the completion of the PHP.

Stage Three: At the end of this six month period the investigators will undertake qualitative interviews with a selection of service users and staff to understand their experience of using the PHP.

The investigators hope to be able to use the results of this pilot study to introduce the use of the PHP into routine care.

DETAILED DESCRIPTION:
The PHP is designed to be very simple to use and there will be 3 versions, 1. paper version, 2. 1 version implemented via the 'IMPARTS' computerised 'tablet' based system that has been separately evaluated (REC Ref 12/SC/0422) and 3. 1 version on an iPad via the Healthlocker system via Mindwaves.

The investigators wish to pilot the use of this PHP in two community teams in the South London and Maudsley (SLaM) Trust. The pilot will be done in three stages.

Stage One: The investigators will undertake an initial qualitative study to refine the process of using the PHP using focus group consultations with staff and service users.

Stage Two: The investigators will then undertake a six month study to evaluate the uptake and use of the PHP. This will involve collecting data on how many people complete the PHP and what actions are taken following the completion of the PHP.

Stage Three: At the end of this six month period the investigators will undertake qualitative interviews with a selection of service users and staff to understand their experience of using the PHP.

The investigators hope to be able to use the results of this pilot study to introduce the use of the PHP into routine care.

ELIGIBILITY:
Inclusion Criteria:

* using one of the community mental health teams recruiting in the study

Exclusion Criteria:

* unable to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in uptake of physical healthcare by service users | Baseline and six months
  Service users will have increased their access to physical healthcare services

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williams J, Sevdalis N, Gaughran F. Evaluation of a Physical health plan for people with psychosis: a protocol for a quality improvement study. Pilot Feasibility Stud. 2019 Jan 15;5:8. doi: 10.1186/s40814-019-0396-7. eCollection 2019. PMID 30675375